CLINICAL TRIAL: NCT04521400
Title: the Investigation Into Beneficial Effects of High-dose Interferon Beta 1-a, Compared to Low-dose Interferon Beta 1-a in Moderate to Severe Covid-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ilad Alavi Darazam, Dr. Ilad Alavi Darazam, MD, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interferon in COVID
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: COVID-19; Interferons; Ritonavir; Lopinavir; Interferon-beta; Antiviral Agents; Anti-Infective Agents; Immunologic Factors
MeSH Terms: conditions — COVID-19 | interventions — Interferon beta-1a; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1 (Experimental): Lopinavir /Ritonavir +high dose Interferon-β 1a
  Interventions: Drug: High dose Interferon-beta 1a; Drug: Lopinavir/Ritonavir
- Arm2 (Experimental): Lopinavir /Ritonavir + Low dose Interferon-β 1a
  Interventions: Drug: Lopinavir/Ritonavir; Drug: Low dose Interferon-beta 1a

INTERVENTIONS:
Drug: High dose Interferon-beta 1a — High dose IFN-β1a (Recigen) (Subcutaneous injections of 88μg (24,000 IU) on days 1, 3, 6)
  Arms: Arm1
Drug: Lopinavir/Ritonavir — Lopinavir/Ritonavir (Kaletra) [IFN-β1a group] (400mg/100 mg twice a day for 10 days
Drug: Low dose Interferon-beta 1a — Low doseIFN-β1a (Recigen) (Subcutaneous injections of 44μg (12,000 IU) on days 1, 3, 6)
  Arms: Arm2

SUMMARY:
The present study is a randomized clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Loghman Hakim Medical Education Center in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

DETAILED DESCRIPTION:
According to previous studies, IFN-β has strong antiviral activity and also has an acceptable safety profile. Based on possible therapeutic effects, we decided to lead an Investigation into Beneficial Effects of high-dose Interferon Beta 1a, Compared to low-dose Interferon Beta 1a (the base therapeutic regimen) in Moderate to Severe COVID-19.

Previous studies demonstrate that IFN-β 1a could be used against some coronaviruses including avium infectious, bronchitis virus, murine hepatitis virus, and SARS- CoV because they are susceptible in vitro or in vivo. In a current study, the efficacy of IFN-β 1a in COVID-19 patients were evaluated, and they found than IFN-β 1a reduced the disease symptoms.

The present study is a randomized clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Loghman Hakim Medical Education Center in Tehran.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* COVID-19 Confirmed Cases (Either RT-PCR or CT Scan Confirmed)
* at least one of the following: radiation contactless body temperature ≥37.5, cough, shortness of breath, nasal congestion/ discharge, myalgia/arthralgia, diarrhea/vomiting, headache or fatigue on admission.
* Time of onset of the symptoms should be acute (Days ≤ 14)
* NEWS2 ≥ 1 on admission (National Early Warning Score 2)

Exclusion Criteria:

* Refusal to participate expressed by patient or legally authorized representative if they are present
* Patients using drugs with potential interaction with Lopinavir/Ritonavir or Interferon-β 1a
* Pregnant or lactating women.
* History of alcohol or drug addiction in the past 5 years.
* Blood ALT/AST levels > 5 times the upper limit of normal on laboratory results.
* The patients who were intubated less than one hours after admission to the hospital

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-20 (Estimated); Primary Completion 2020-09-04 (Estimated); Study Completion 2020-09-11 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | From date of randomization until 14 days later
  Improvement of two points on a seven-category ordinal scale (recommended by the World Health Organization: Coronavirus disease (COVID-2019) R&D. Geneva: World Health Organization) or discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Mortality | From date of randomization until 14 days later
  If the patient dies, we have reached an outcome
SpO2 Improvement | Days 1, 2, 3, 4, 5, 6, 7 and 14
  Pulse-oxymetry
Incidence of new mechanical ventilation use | From date of randomization until 14 days later
Duration of hospitalization | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 14 days
Cumulative incidence of serious adverse events | Days 1, 2, 3, 4, 5, 6, 7 and 14
  With the incidence of any serious adverse effects, the outcome has happened

CONTACTS AND LOCATIONS:
Overall Officials: Ilad Alavi Darazam, M.D, Study Chair — Shahid Beheshti University of Medical Sciences; Firouze Hatami, M.D, Principal Investigator — Shahid Beheshti University of Medical Sciences; Mohammad Mahdi Rabiei, M.D, Principal Investigator — Shahid Beheshti University of Medical Sciences; Omid Moradi, Principal Investigator — Shahid Beheshti University of Medical Sciences; Behnam Rahimi, M.D, Principal Investigator — Shahid Beheshti University of Medical Sciences; Shervin Shokouhi, M.D, Study Director — Shahid Beheshti University of Medical Sciences; Mohammad Reza Hajesmaeili, M.D, Principal Investigator — Shahid Beheshti University of Medical Sciences; Minoosh Shabani, M.D, Principal Investigator — Shahid Beheshti University of Medical Sciences; Seyed Sina Naghibi Irvani, M.D, Principal Investigator — Shahid Beheshti University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yan R, Zhang Y, Li Y, Xia L, Guo Y, Zhou Q. Structural basis for the recognition of SARS-CoV-2 by full-length human ACE2. Science. 2020 Mar 27;367(6485):1444-1448. doi: 10.1126/science.abb2762. Epub 2020 Mar 4. PMID 32132184
- [Background] Ou X, Liu Y, Lei X, Li P, Mi D, Ren L, Guo L, Guo R, Chen T, Hu J, Xiang Z, Mu Z, Chen X, Chen J, Hu K, Jin Q, Wang J, Qian Z. Characterization of spike glycoprotein of SARS-CoV-2 on virus entry and its immune cross-reactivity with SARS-CoV. Nat Commun. 2020 Mar 27;11(1):1620. doi: 10.1038/s41467-020-15562-9. PMID 32221306
- [Background] Zheng HY, Zhang M, Yang CX, Zhang N, Wang XC, Yang XP, Dong XQ, Zheng YT. Elevated exhaustion levels and reduced functional diversity of T cells in peripheral blood may predict severe progression in COVID-19 patients. Cell Mol Immunol. 2020 May;17(5):541-543. doi: 10.1038/s41423-020-0401-3. Epub 2020 Mar 17. No abstract available. PMID 32203186
- [Background] Wang BX, Fish EN. Global virus outbreaks: Interferons as 1st responders. Semin Immunol. 2019 Jun;43:101300. doi: 10.1016/j.smim.2019.101300. PMID 31771760
- [Background] Hung IF, Lung KC, Tso EY, Liu R, Chung TW, Chu MY, Ng YY, Lo J, Chan J, Tam AR, Shum HP, Chan V, Wu AK, Sin KM, Leung WS, Law WL, Lung DC, Sin S, Yeung P, Yip CC, Zhang RR, Fung AY, Yan EY, Leung KH, Ip JD, Chu AW, Chan WM, Ng AC, Lee R, Fung K, Yeung A, Wu TC, Chan JW, Yan WW, Chan WM, Chan JF, Lie AK, Tsang OT, Cheng VC, Que TL, Lau CS, Chan KH, To KK, Yuen KY. Triple combination of interferon beta-1b, lopinavir-ritonavir, and ribavirin in the treatment of patients admitted to hospital with COVID-19: an open-label, randomised, phase 2 trial. Lancet. 2020 May 30;395(10238):1695-1704. doi: 10.1016/S0140-6736(20)31042-4. Epub 2020 May 10. PMID 32401715
- [Background] Hensley LE, Fritz LE, Jahrling PB, Karp CL, Huggins JW, Geisbert TW. Interferon-beta 1a and SARS coronavirus replication. Emerg Infect Dis. 2004 Feb;10(2):317-9. doi: 10.3201/eid1002.030482. PMID 15030704
- [Background] Dastan F, Nadji SA, Saffaei A, Marjani M, Moniri A, Jamaati H, Hashemian SM, Baghaei P, Abedini A, Varahram M, Yousefian S, Tabarsi P. Subcutaneous administration of interferon beta-1a for COVID-19: A non-controlled prospective trial. Int Immunopharmacol. 2020 Aug;85:106688. doi: 10.1016/j.intimp.2020.106688. Epub 2020 Jun 7. PMID 32544867
- [Derived] Alavi Darazam I, Hatami F, Mahdi Rabiei M, Amin Pourhoseingholi M, Shabani M, Shokouhi S, Mardani M, Moradi O, Javandoust Gharehbagh F, Mirtalaee N, Negahban H, Amirdosara M, Zangi M, Hajiesmaeili M, Kazempour M, Shafigh N. An investigation into the beneficial effects of high-dose interferon beta 1-a, compared to low-dose interferon beta 1-a in severe COVID-19: The COVIFERON II randomized controlled trial. Int Immunopharmacol. 2021 Oct;99:107916. doi: 10.1016/j.intimp.2021.107916. Epub 2021 Jun 29. PMID 34224994
- [Derived] Alavi Darazam I, Hatami F, Rabiei MM, Pourhoseingholi MA, Moradi O, Shokouhi S, Hajesmaeili MR, Shabani M, Irvani SSN. An investigation into the beneficial effects of high-dose interferon beta 1-a, compared to low-dose interferon beta 1-a (the base therapeutic regimen) in moderate to severe COVID-19: A structured summary of a study protocol for a randomized controlled l trial. Trials. 2020 Oct 26;21(1):880. doi: 10.1186/s13063-020-04812-2. PMID 33106183